CLINICAL TRIAL: NCT02766855
Title: Efficacy of Topical Cysteamine in Nephropathic Cyctinosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Eye Center and The Eye Foundation for Research in Ophthalmology (Other)
Responsible Party: Principal Investigator, Samir S. Shoughy, MD, FRCS (Glasg.), Ophthamolgist, uveitis, Cornea & External Eye Disease, The Eye Center and The Eye Foundation for Research in Ophthalmology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TEC C123
Record Dates: First submitted 2016-04-12; First posted 2016-05-10 (Estimated); Last update posted 2016-05-10 (Estimated); Status verified 2016-05

CONDITIONS: Nephropathic Cyctinosis; Corneal Cystine Crystals
Keywords: cysteamine; nephropathic cystinosis; cystine crystals
MeSH Terms: conditions — Cystinosis | interventions — Cysteamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- cysteamine eye drops (Experimental): Patients used cysteamine eye drops every 2 hours while awake to both eyes.
  Interventions: Drug: Cysteamine

INTERVENTIONS:
Drug: Cysteamine — Patients were asked to use topical cysteamine 0.55% eye drops every 2 hours while awake to both eyes.

SUMMARY:
The aim of this study is to evaluate the efficacy of topical cysteamine eye drops in the treatment of corneal cystine crystals deposits in patients with nephropathic cystinosis.

DETAILED DESCRIPTION:
A total of 26 patients with nephropathic cystinosis were included in this prospective study. Patients were evaluated for improvement of corneal cysteine deposits crystals and photophobia following treatment with topical 0.55% cysteamine eye drops.

ELIGIBILITY:
Inclusion Criteria:

* patients with confirmed diagnosis of nephropathic cystinosis
* leucocyte cystine concentration level of more than 2.0 nmol half-cystine/ mg protein
* clinical evidence of tissue deposition of cystine and tissue damage due to cystinosis

Exclusion Criteria:

* Allergy to cysteamine

Ages: 8 Months to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 26 (Actual)
Dates: Start 2004-01; Primary Completion 2012-12 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Number of participants with improvement of photophobia, corneal cystine crystals and visual acuity following treatment with topical cysteamine 0.55% eye drops in patients with nephropathic cystinosis. | Photophobia, slit lamp assessment of corneal cystine crystals and visual acuity are recorded pretreatment, on each monthly visit up to 48 months.
  Patients had a baseline ophthalmic examination before initiation of topical cysteamine 0.55% eye drops and subsequent monthly follow up exams. The following parameters were recorded pretreatment, on each monthly visit and post treatment at last follow up visit: photophobia, slit lamp assessment of corneal cystine crystals and visual acuity. Photophobia was classified as grade 0 (none) for no photophobia, grade 1 (mild) for photophobia in bright light, grade 2 (moderate) for photophobia in room light and grade 3 (severe) for photophobia in dim light. Corneal cystine crystals were graded as Grade 0 = None, Grade 1 = 1-10 crystals/mm, Grade 2 = 11- 50 crystals/mm, Grade 3 = more than 50 crystals/mm. The level of cystine in the corneal layers was recorded and the location whether peripheral or central was also identified. Visual acuity was measured by Snellen chart at 20 feet with best distance correction.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Al-Hemidan A, Shoughy SS, Kozak I, Tabbara KF. Efficacy of topical cysteamine in nephropathic cystinosis. Br J Ophthalmol. 2017 Sep;101(9):1234-1237. doi: 10.1136/bjophthalmol-2016-309278. Epub 2017 Jan 5. PMID 28057644